CLINICAL TRIAL: NCT04697641
Title: Efficacy of Helicobacter Pylori Eradication on Symptoms of Functional Dyspepsia - A Randomised Controlled Trial
Brief Title: Helicobacter Pylori Eradication in Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Piyush Ranjan, Professor, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/07/17/1202
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Dyspepsia; Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Functional Dyspepsia; Triple Drug Regimen; Global Overall Scale; Epigastric Pain Syndrome
MeSH Terms: conditions — Dyspepsia | interventions — Clarithromycin; Amoxicillin; Pantoprazole; levosulpiride; Z 338; itopride

STUDY DESIGN:
Intervention Model Description: Two study groups receiving two different treatment strategies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Helicobacter pylori eradication therapy Group (Experimental): Patients with Functional Dyspepsia receiving two week course of triple drug regimen for H pylori eradication followed by six weeks of proton pump inhibitors
  Interventions: Drug: Clarithromycin 500mg; Drug: Amoxicillin 1000 MG; Drug: Pantoprazole 40mg
- Symptomatic treatment group (Active Comparator): Patients with Functional Dyspepsia receiving symptomatic therapy with proton pump inhibitors or gastric prokinetics
  Interventions: Drug: Pantoprazole 40mg; Drug: Levosulpiride; Drug: Acotiamide; Drug: Itopride

INTERVENTIONS:
Drug: Clarithromycin 500mg — Clarithromycin 500 mg twice a day for two weeks
  Arms: Helicobacter pylori eradication therapy Group
Drug: Amoxicillin 1000 MG — Amoxicillin 1000mg twice a day for two weeks
  Arms: Helicobacter pylori eradication therapy Group
Drug: Pantoprazole 40mg — Pantoprazole 40 mg or equivalent for eight weeks
Drug: Levosulpiride — Levosulpiride 25 mg as and when required before meals
  Arms: Symptomatic treatment group
Drug: Acotiamide — Acotiamide 100mg as when required before meals
  Arms: Symptomatic treatment group
Drug: Itopride — Itopride 50mg as when required before meals
  Arms: Symptomatic treatment group

SUMMARY:
This study is designed to study benefit of eradicating Helicobacter Pylori in patients with functional dyspepsia as compared to symptomatic treatment only. Helicobacter pylori positive patients with Functional Dyspepsia will be divided into two study groups, one will receive Helicobacter pylori eradication therapy and other will receive symptomatic treatment. Symptom relief based on Likert scale will be compared in both groups.

DETAILED DESCRIPTION:
Functional dyspepsia (FD), is a common problem with many associations. About 50% of the patients with FD have coexistent Helicobacter pylori (HP) associated gastritis.

Many investigators have tried to treat FD by means of eradication of HP infection. Different studies have reported various estimates of association between HP eradication and improvement of dyspeptic symptoms, and whether eradication of HP infection improves dyspeptic symptoms in patients with FD remains controversial because of scarcity of large randomised controlled studies, and great heterogeneity in study designs. Also, antibiotic use or misuse is widely prevalent; the resultant high frequency of antibiotic resistance implies that treatment regimens for HP eradication may not be effective. On this background, the investigators propose to conduct a large tertiary centre based study to find the effect of eradicating HP on the symptoms of FD. Secondarily, the investigators also propose to look for prevalence of HP in FD and recurrence rate of HP infection at 6 month follow up after the eradication therapy.

The investigators hypothesise that HP eradication is superior to Standard of care symptomatic management in treating symptoms of FD.

Primary Objectives:

• To study the effect of HP eradication on symptom profile of Functional Dyspepsia.

Secondary Objectives:

* To determine the prevalence of HP infection in patients with Functional Dyspepsia (FD).
* To study the efficacy of HP eradication therapy.
* To study the recurrence rate of HP infection and symptom relief at 6 months follow up after completion of treatment.

Study Centre: The study will be carried out at Sir Ganga Ram Hospital, New Delhi.

Study Design: This will be open label randomised controlled study. Study Duration: Study will be conducted from 1st September 2017 to 31st May 2019, with patient recruitment till 30th November 2018. Study would start after obtaining requisite Ethical Clearance from Institutional Ethical Committee.

Patients to be enrolled: Consecutive patients of Functional Dyspepsia, according to ROME-IV criteria, who attend the gastroenterology Out patient departement at our centre.

Patient selection:

Patients who will seek medical care for dyspeptic symptoms present for at least three months and those who have no history of peptic ulcer disease or gastroesophageal disease or previous treatment for HP will be eligible for the study.

Inclusion and exclusion criteria will be applied and final study sample will be calculated.

Blood investigations like complete hemogram, liver function tests, renal function tests, TSH, urine analysis, fasting and post prandial blood sugar levels, HbA1c if required and an ultrasound abdomen will be done. Those with uncontrolled diabetes mellitus (HbA1c>9mmol/mol) and uncontrolled thyroid status (TSH>10mIU/l or <0.5mIU/L) will be excluded from the study.

Other participants will be subjected to upper GI endoscopy and those with normal Upper GI Endoscopy will fulfil the ROME IV criteria of FD. A RUT and HP stool Ag test will be done for them. A positive result for both the test will be considered as HP positive. This will be used to find the prevalence of HP in FD. Those with a single positive test will be considered negative.

HP negative FD patients will receive the standard of care treatment.

Symptom Assessment:

The Global Overall Symptom (GOS) scale will be used for symptom assessment. The symptoms are reported on a seven point Likert Scale ranging from 1 = no problem to 7 = very severe problem. The GOS score is self-reported by the patient over a retrospective period of 28 days. Those with moderate to high intensity (>2 on Likert Scale) of symptoms will be included in the study.

Patients will also be asked to rate the severity of 10 specific upper GI symptoms [specific symptom subtypes (SSS)] using the same 7-point Likert scale as for the GOS scale: epigastric pain, epigastric discomfort, heartburn, acid regurgitation, upper abdominal bloating, excessive belching, nausea, early satiety, postprandial fullness and other epigastric symptoms. Participants will be divided into two symptom subgroups- Epigastric Pain Syndrome (EPS)- for first four symptoms on GOS; and Post Prandial Distress Syndrome (PDS)- for last six symptoms on GOS.

Randomisation and Intervention:

H.pylori positive FD patients will be randomised to two arms based on computer generated randomisation.

* One arm will receive H.pylori eradication therapy in the form of fourteen days of Tab.Clarithromycin 500 mg twice a day + Tab.Amoxicillin 1000mg twice a day+ Tab. Pantoprazole 40mg twice a day followed by six more weeks of Tab.Pantoprazole 40mg once daily.
* Other arm would receive the standard of care treatment for FD, i.e, proton pump inhibitors for eight weeks in case EPS and prokinetics as when required for patients with PDS.

Follow up:

The first follow up will be four weeks after completion of eight week treatment. On this follow up, GOS will be administered and rating of 0 or 1 on the Likert Scale will be considered as symptom relief and treatment success. H.pylori Stool Ag test will be done and positive H.pylori Stool Ag test will be taken as failure of H.pylori eradication.

The second follow up will be after six months of completion of eight week treatment. GOS and SSS will be asked and H.pylori Stool Ag testing will be repeated. Participants may receive medications for symptom relief over these six months and a note will be made about the treatment in their diary. Symptoms hampering their routine daily activities will be taken as failure of symptom relief.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients fulfilling the ROME-IV criteria of Functional Dyspepsia
* Signed informed consent.

Exclusion Criteria:

* Pregnant and lactating females
* Patients with predominant symptoms of heartburn or irritable bowel syndrome; alarm symptoms; history of peptic ulcer, upper gastrointestinal tract surgery, or biliary colic
* Previous treatment for eradication of H pylori.
* Known allergies to study medication or alcohol or drug abuse.
* Use of antibiotics or bismuth during the 4 weeks before enrolment, proton pump inhibitors during the 2 weeks before enrolment, or treatment with histamine-2 receptor blockers in the week before enrolment will not be permitted.
* Patients unable to answer the study questionnaires.
* Patients unwilling or unable to provide consent.
* Patient on HIV/AIDS medications, blood thinners, clopidogrel, cyclosporine, digoxin, iron supplements, fluconazole or ketoconazole, probenecid, rifabutin, sildenafil, tacrolimus, theophylline, sulfa drugs, cholesterol-lowering medicines, heart rhythm medications, sedatives, seizure medications, or tetracycline antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Treatment Success | Six months after the completion of intervention
  Treatment success defined as absence of symptoms or minimal symptoms (GOS score <3) with GOS reduction by at least 2, 6 months after treatment.

SECONDARY OUTCOMES:
Prevalence of Helicobacter pylori infection in Functional Dyspepsia | At enrolment
  Proportion of Helicobacter pylori positive patients with Functional Dyspepsia
Efficacy of Helicobacter pylori eradication therapy | Four weeks after the completion of intervention
  Efficacy of Helicobacter pylori eradication therapy defined as stool HP Ag negative at 4 weeks after treatment.
Rate of Helicobacter pylori reinfection | Six months after the completion of intervention
  Rate of Helicobacter pylori reinfection defined as Stool HP Ag positivity at 6 months in those who were negative at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology & Hepatology, Sir Ganga Ram Hospital, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Padole P, Ranjan P, Sachdeva M, Kumar M. Role of Helicobacter pylori eradication in patients with functional dyspepsia. Indian J Gastroenterol. 2021 Oct;40(5):492-501. doi: 10.1007/s12664-021-01195-3. Epub 2021 Oct 27. PMID 34708338